CLINICAL TRIAL: NCT03149705
Title: CoHort of Patients to Identify Biological and Imaging markerS of CardiovascUlar Outcomes in Stroke.
Brief Title: Cohort of Ischemic STROKE Patients
Acronym: HIBISCUSSTROKE
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0323
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke, stroke, bio-collection, Imaging markers, biomarkers, clinical outcomes
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In usual care of patients admitted for ischemic STROKE at Pierre Wertheimer Hospital, blood samples were taken on admission in the neurovascular unit (H0), 6h, 24h and 48h after reperfusion , and during the 3 month clinical visit.
  For the constitution of the serum bank of Hibiscus-STROKE cohort, extra tubes are collected at the same time as the blood tests done routinely.
  These additional samples will be centrifuged and treated to form a collection of biological samples of total serum and plasma and blood stored at the Biological Resource Center of HCL Neurobiotec at -80 ° C (DC- 2008-72, AC-2013-1867 certified NFS96900 FR13-018140).
Oversight: Data Monitoring Committee: No

SUMMARY:
Ischemic stroke is the first cause of acquired disability of the adult, the second cause of dementia and the third cause of death in the industrialized countries, what constitutes à major public health issue. Stroke is characterized by a cerebral parenchymal lesion due to an ischemic mechanism (85% of the cases) or hemorrhagic mechanism (15%). For a long time, the only approved treatment was the intravenous thrombolysis (rt-PA). Recently, thrombectomy has proven its superiority in this pathology.

Cohorts of patients with stroke are rare but can be very valuable by their clinical, laboratory and imaging well documented. They are the source of new hypotheses for research or interventions as well as the quality of care assessment tool.

The main objective of this project is to identify new markers: biological and imaging, treatment response and prognosis after ischemic stroke.

Secondary objectives of the HIBISCUS-STROKE cohort are to establish a clinical database, completed by biological samples and by imaging data that can be used in the following areas:

* Descriptive epidemiology of ischemic stroke and cerebral reperfusion,
* Pharmacoepidemiology and treatments observatory: safety, efficacy, indication of treatment in real life, costs
* Assessment of the long-term effect of the treatment on the occurrence of disability, stroke recurrence and death,
* Quality of life and personal, familial, professional and social consequences of stroke,
* Research of new diagnostic and prognostic biomarkers,
* Research projects.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Ischemic Stroke confirmed by MRI
* Proximal arterial occlusion (ICA or M1)
* Eligible for thrombolysis and/or thrombectomy

Exclusion Criteria:

* Patients residing> 50 km from the Pierre Wertheimer Hospital (Lyon, France)
* Inability to perform the first sample (H0)
* Patient with progressive or uncontrolled cancer.
* Refusal to participate in the study or to sign the consent
* Lack of medical social coverage
* Deprivation of civil rights

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-10-13 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Degree of disability (mRS Score) | 5 years
  Degree of disability: modified Rankin Score

SECONDARY OUTCOMES:
infarct size | day 6
  cerebral infarct size on MRI
Hemorrhagic transformation | 24 hours
  Hemorrhagic transformation (ECASS scale) on imaging (CT or MRI)
Neurological deficit | up to 5 years
  Neurological deficit NIH stroke Scale
Quality of life | up to 5 years
  QOL questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital neurologique Pierre Wertheimer (Lyon), Bron, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bani-Sadr A, Hermier M, de Bourguignon C, Mechtouff L, Eker OF, Cappucci M, Tommasino E, Martin A, Cho TH, Derex L, Nighoghossian N, Berthezene Y. Oxygen Extraction Fraction Mapping on Admission Magnetic Resonance Imaging May Predict Recovery of Hyperacute Ischemic Brain Lesions After Successful Thrombectomy: A Retrospective Observational Study. Stroke. 2024 Nov;55(11):2685-2693. doi: 10.1161/STROKEAHA.124.047311. Epub 2024 Oct 11. PMID 39391984